CLINICAL TRIAL: NCT04084665
Title: A Pilot Study to Examine Safety, Activity and Biomarkers in Participants With Hidradenitis Suppurativa Receiving a Previously Tested Subcutaneous Dose of Anti-IL-23 Monoclonal Antibody Guselkumab.
Brief Title: Biomarkers in Participants With Hidradenitis Suppurativa Receiving Guselkumab.
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Rockefeller University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JFR-0992
Record Dates: First submitted 2019-09-09; First posted 2019-09-10 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — guselkumab

STUDY DESIGN:
Intervention Model Description: Single Arm Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Guselkumab 200mg q4 weekly
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab

SUMMARY:
Hidradenitis Suppurativa (HS) is a severe, chronic debilitating disease with a variable and incomplete response to current treatments. Existing immunological studies have found dysregulation in the TH17:Treg axis with an increase in inflammatory mediators including TNFalpha, IL-17 IL-23 (amongst others) in lesional skin. Multiple cell typesincluding CD4+ cells, dendritic cells and macrophages infiltrate active lesions of HS and produce this major contribution from the Th17 axis.

One of the main barriers to the development of novel and effective treatments for HS is the lack of biomarker(s) of disease activity, as well as our incomplete understanding of the pathogenesis of this disease. Given the pronounced contribution of Th17 pathway (including interleukin-23) in the inflammation in HS, further investigation into the role of this axis in the pathogenicity of HS is essential. Guselkumab is a fully human interluekin-23 antagonist, FDA approved for the treatment of moderate to severe psoriasis in participants 18 years and over. Guselkumab is a novel potential therapy.

DETAILED DESCRIPTION:
Hidradenitis Suppurativa (HS) is a severe, chronic debilitating disease with a variable and incomplete response to current treatments. Existing immunological studies have found dysregulation in the TH17:Treg axis with an increase in inflammatory mediators including TNFalpha, IL-17 IL-23 (amongst others) in lesional skin. Multiple cell typesincluding CD4+ cells, dendritic cells and macrophages infiltrate active lesions of HS and produce this major contribution from the Th17 axis.

One of the main barriers to the development of novel and effective treatments for HS is the lack of biomarker(s) of disease activity, as well as our incomplete understanding of the pathogenesis of this disease. Markers such as C- Reactive Protein, IL-6, soluble IL-2 receptor, S100A8/9, lipocalin-2 and the neutrophil/lymphocyte rati7 have been proposed as potential biomarkers but lack high specificity and correlation with disease severity. Given the pronounced contribution of Th17 pathway (including interleukin-23) in the inflammation in HS, further investigation into the role of this axis in the pathogenicity of HS is essential. Guselkumab is a fully human interluekin-23 antagonist, FDA approved for the treatment of moderate to severe psoriasis in participants 18 years and over. Guselkumab is a novel potential therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe Hidradenitis Suppurativa (HS) for at least 1 year (365 days) prior to the baseline visit as determined by the investigator through participant interview and/or review of medical history
* Have HS lesions present in at least 2 distinct anatomical areas
* Had an inadequate response to an adequate course of appropriate oral antibiotics for treatment of HS (or demonstrated intolerance to, or had contraindications to oral antibiotic treatment of their HS
* Have a total abscess and inflammatory nodule (AN) count greater than or equal to 3 at the screening and baseline visit
* Must agree with daily use (throughout the study of one of the following over the counter treatments to body areas affected with HS lesions: either soap and water, a topical antiseptic was containing chlorhexidine gluconate, triclosan or benzoyl peroxide, or a dilute bleach bath.

Exclusion Criteria:

* HIV Positive
* Active Hepatitis B or C Infection
* Pregnant or Breastfeeding
* No concurrent use of any systemic antibiotics/retinoids/immunosuppressants (require washout period of 5 half lives)
* Any medical, psychological or social condition that, in the opinion of the investigator would jeopardize the health or well being of the participant during any study procedures or integrity of the data
* Has a draining fistula count greater than 20 at baseline visit Any other active skin disease (bacterial fungal or viral infection) that could have interfered with the assessment of HS

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Biomarkers at Week 12 | Week 12 compared with baseline (Week 0).
  Change in lesional tissue levels of IL-17A, IL-17C, IL-17F and IL-23, measured in pg/mL
Biomarkers at Week 24 | Week 24 compared with baseline (Week 0).
  Primary Outcomes would be the change in lesional tissue levels of IL-17A, IL-17C, IL-17F and IL-23 measured in pg/mL measured in pg/mL
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 0 to Week 24
  Incidence of Grade 2/3 adverse events during the study

SECONDARY OUTCOMES:
Clinical Response at Week 12 (as measured by HiSCR) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by the HiSCR (Hidradenitis Suppurativa Clinical Response) Defined as a greater than or equal to 50% reduction in inflammatory lesion count (abscesses plus inflammatory nodules), and no increase in abscesses or draining fistulas at Week 12 when compared with baseline
Clinical Response at Week 12 (as measured by modified Sartorius Score) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by the modified Sartorius Score as follows: Sum of separate scoring for each affected area using the data recorded as follows: a) 3 points per anatomical region involved; b) 6 points for each fistula and 1 point for each nodule or abscess; c) 1 point when the longest distance between two relevant lesions in each affected area is <5 cm; 3 points when it is 5-10 cm; and 9 points when it is >10 cm; d) 9 points when there is no clear separation of lesions from adjacent normal skin and 0 points when there is.
Clinical Response at Week 12 (as measured by IHS4) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by IHS4 (International Hidradenitis Suppurativa Severity Score) using the scoring system as follows: Total= (Number of nodules x1) + (Number of abscesses x2) + (Number of draining sinuses/fistulae x4)
Clinical Response at Week 24 (as measured by HiSCR) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by the HiSCR (Hidradenitis Suppurativa Clinical Response) Defined as a greater than or equal to 50% reduction in inflammatory lesion count (abscesses plus inflammatory nodules), and no increase in abscesses or draining fistulas at Week 24 when compared with baseline
Clinical Response at Week 24 (as measured by modified Sartorius Score) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by the modified Sartorius Score as follows: Sum of separate scoring for each affected area using the data recorded as follows: a) 3 points per anatomical region involved; b) 6 points for each fistula and 1 point for each nodule or abscess; c) 1 point when the longest distance between two relevant lesions in each affected area is <5 cm; 3 points when it is 5-10 cm; and 9 points when it is >10 cm; d) 9 points when there is no clear separation of lesions from adjacent normal skin and 0 points when there is.
Clinical Response at Week 24 (as measured by IHS4) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by IHS4 (International Hidradenitis Suppurativa Severity Score) using the scoring system as follows: Total= (Number of nodules x1) + (Number of abscesses x2) + (Number of draining sinuses/fistulae x4)

CONTACTS AND LOCATIONS:
Overall Officials: John W Frew, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller Unviersity, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No